CLINICAL TRIAL: NCT05145894
Title: Differentiation of Asthma/COPD Exacerbation and Stable State Using Automated Lung Sound Analysis With LungPass Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Healthy Networks (Industry)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: № 4-3/YH-2056/LP05
Record Dates: First submitted 2021-10-21; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Asthma; COPD
Keywords: Lung sound analysis; Asthma Exacerbation; COPD Exacerbation
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma: Asthma patients aged 3 years and older with confirmed asthma diagnosis treated by a monotherapy ICS or ICS plus LABA or other controllers and presenting with moderate or severe disease exacerbation
  Interventions: Device: Lung auscultation with LungPass device (electronic auscultation)
- COPD: COPD patients aged 40 years and older with confirmed COPD diagnosis treated by a monotherapy long-acting muscarinic antagonist (LAMA), or LAMA plus long acting beta2-agonist (LABA), or inhaled corticosteroid (ICS) plus LABA, or LAMA plus LABA plus ICS and presenting with moderate or severe disease exacerbation
  Interventions: Device: Lung auscultation with LungPass device (electronic auscultation)

INTERVENTIONS:
Device: Lung auscultation with LungPass device (electronic auscultation) — Lung auscultation with electronic stethoscope

SUMMARY:
This observational study evaluates whether lung sound analysis with LungPass device can be used to differentiate exacerbation and stable state asthma and COPD.

DETAILED DESCRIPTION:
This is a prospective observational study comprised patients with moderate or severe COPD or asthma exacerbation in primary care settings. Patients will be examined twice - during an exacerbation of the disease and in a stable phase. Patients will undergo routine clinical examination including lung auscultation with conventional stethoscope and LungPass device. Moreover, symptoms and anamnesis data, results of symptoms questionnaires (CAT for COPD and ACQ-5 for asthma), result of diagnostic questionnaire from the LungPass App, spirometry data, serum procalcitonin (for COPD patients), C-reactive protein, white blood cell count and blood eosinophil count, results of sputum cytology examination, Х-ray results (if carried out according to indications) will be collected.

ELIGIBILITY:
Inclusion Criteria:

For COPD patients:

* Patients able and willing to sign an informed consent to participate in the study;
* Patient is aged 40 years or older with a smoking history of ≥10 pack years;
* Patients with COPD confirmed previously by a detailed medical history and examination;
* Patients presenting with moderate or severe exacerbation of chronic obstructive pulmonary disease.
* Patient is treated by a monotherapy long-acting muscarinic antagonist (LAMA), or LAMA plus long acting beta2-agonist (LABA), or inhaled corticosteroid (ICS) plus LABA, or LAMA plus LABA plus ICS.

For asthma patients:

* Patients able and willing to sign an informed consent to participate in the study;
* Patient is aged 3 years or older;
* Patients with asthma confirmed previously by a detailed medical history and examination;
* Patients presenting with moderate or severe exacerbation of asthma;
* Patient is treated by a monotherapy ICS or ICS plus LABA or other controllers.

Exclusion Criteria:

* Age up to 3 years for asthma patients and up to 40 years for COPD patients;
* Patient refusal to participate in the study;
* Patients with subcutaneous emphysema, with damaged skin on the surface of the chest, with drainage in the pleural space, patients undergoing mechanical ventilation;
* Patients with asthma-COPD overlap or presence of other known chronic lung conditions such tuberculosis, cystic fibrosis or clinically significant bronchiectasis;
* Mental illness, other known acute diseases or known chronic decompensated diseases, such as a known active malignancy or severe heart failure, other known ongoing infection.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — for COPD: 40 years or older for asthma: 3 years or older
Study Population: Patients will be recruited upon presentation with a moderate or severe COPD or asthma exacerbation in primary care settings.
  It is planned to recruit 100 patients with asthma and 100 patients with COPD at the initial study stage. The final calculation of the sample size will be carried out after receiving the preliminary results of the study. After that, the sample size will be adjusted.
  Patients will be examined twice - during an exacerbation of the disease and in a stable phase.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of asthma exacerbation detection by lung sounds | 30.09.2021-30.09.2022
  Accuracy of identifying acute exacerbation of asthma by abnormal lung sounds detected with LungPass device.
Accuracy of COPD exacerbation detection by lung sounds | 30.09.2021-30.09.2022
  Accuracy of identifying acute exacerbation of chronic obstructive pulmonary disease by abnormal lung sounds detected with LungPass device.

SECONDARY OUTCOMES:
Lung sounds and symptoms correlation in patients with asthma exacerbation | 30.09.2021-30.09.2022
  Correlation between the presence of pathological pulmonary sounds and the presence of symptoms of asthma exacerbation
Lung sounds and symptoms correlation in patients with COPD exacerbation | 30.09.2021-30.09.2022
  Correlation between the presence of pathological pulmonary sounds and the presence of symptoms of COPD exacerbation

OTHER OUTCOMES:
Accuracy of asthma exacerbation detection by LungPass App output | 30.09.2021-30.09.2022
  Аccuracy of identifying acute exacerbation of chronic obstructive pulmonary disease and asthma by final LungPass App output which based on abnormal lung sounds detected with LungPass device together with symptoms collected using a questionnaire in the LungPass app*.
  * Final LungPass App output is possible patient condition (asthma/asthma exacerbation, COPD/COPD exacerbation, bronchitis, pneumonia, etc)
Accuracy of COPD exacerbation detection by LungPass App output | 30.09.2021-30.09.2022
  Аccuracy of identifying acute exacerbation of chronic obstructive pulmonary disease by final LungPass App output which based on abnormal lung sounds detected with LungPass device together with symptoms collected using a questionnaire in the LungPass app*.
  * Final LungPass App output is possible patient condition (asthma/asthma exacerbation, COPD/COPD exacerbation, bronchitis, pneumonia, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Binetskaya, Study Director — CEO
Locations (1):
- Minsk Clinical Phthisiopulmonology Center, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided